CLINICAL TRIAL: NCT03428763
Title: ELECTOR Treat-to-target Via Home-based Disease Activity Monitoring of Patients With Rheumatoid Arthritis: A 6 Months Multicentre, eHealth Randomised, Non-blinded, Parallel-group, Superiority Trial
Brief Title: ELECTOR Treat-to-target Via Home-based Disease Activity Monitoring of Patients With Rheumatoid Arthritis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Technical problems with POC
Sponsor: Frederiksberg University Hospital (Other)
Responsible Party: Principal Investigator, Henning Bliddal, Head of the Parker Institute, Frederiksberg University Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: APPI-100.02
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2025-02-27 (Actual); Status verified 2020-09

CONDITIONS: Arthritis, Rheumatoid; Telerehabilitation
Keywords: Arthritis, Rheumatoid; Telerehabilitation; controlled randomised trial
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Intervention Model Description: The current trial is designed to assess whether the effectiveness of home-based disease activity monitoring via a home-based (eHealth) intervention is superior to standard clinical disease activity assessment in obtaining and maintaining a low(er) disease activity in patients with RA.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Homebased disease monitoring (eHealth) (Experimental): Participants allocated to the intervention group will be trained in self-monitoring of their RA
  Interventions: Device: Homebased disease monitoring (eHealth)
- Standard clinical disease monitoring (Active Comparator): Those allocated to the control arm of the study will continue usual clinical care (i.e. they will not self-monitor or have access to the eHealth solution). No other medication changes will be mandated and participating investigators will be asked to manage all other care according usual clinical practice. Individuals in the control group will not be given the option to self-monitor.
  Interventions: Other: Standard clinical disease monitoring

INTERVENTIONS:
Device: Homebased disease monitoring (eHealth) — Participants allocated to the intervention group will be trained in self-monitoring (assessment of tender of swollen joints). Further they will be instructed in using a point-of-care CRP-measuring device to measure blood concentrations of C-reactive protein at their home, and to submit the self-monitoring results on a dedicated internet platform. These procedures represent a "virtual visit".
  The participants are instructed to have "virtual visit" (self-monitoring) every month from allocation. The scheduled "virtual visits" include
  * Joint score by the patient
  * Patient global disease activity measured on a 0-100 mm visual analogue scale.
  * CRP measurement on home-based device Based on the submitted data a DAS28-CRP is calculated and recorded in the eCRF.
  Arms: Homebased disease monitoring (eHealth)
Other: Standard clinical disease monitoring — Those allocated to the control arm of the study will continue usual clinical care (i.e. they will not self-monitor or have access to the eHealth solution). No other medication changes will be mandated and participating investigators will be asked to manage all other care according usual clinical practice. Individuals in the control group will not be given the option to self-monitor.
  Arms: Standard clinical disease monitoring

SUMMARY:
The aim of this study is to explore whether the effectiveness of home-based disease activity monitoring via a home-based (eHealth) intervention is superior to standard clinical disease activity assessment in obtaining and maintaining a low(er) disease activity in patients with rheumatoid arthritis (RA).

DETAILED DESCRIPTION:
The aim of RA therapy is to reduce disease activity, joint destruction, symptoms, and disability. The prevailing therapeutic approach is an aggressive pharmacological disease control, with readily available conventional synthetic disease modifying anti-rheumatic drugs (csDMARDs) in first line. The csDMARDs goes a long way towards reductions in disease activity, symptoms, and disability. However, if satisfactory disease control is not achieved by csDMARDS, addition of biologic medicines can be necessary.

With the efficacy of all these pharmacological options and the current view on "Treat-to-Target" (T2T), RA patients should have excellent prospects. However, despite the evidence to support a T2T strategy it is anticipated that many patients across various countries in Europe have active disease and suffer from increasing disability; this might be a consequence of bad access to optimal care, as well as possibly a lack of reimbursement of biological agents. Currently, the proposed T2T strategies are managed in the clinic by physicians, nurses and biometricians, which is expensive and time consuming for both patients and health care professionals (HCPs).

Telemonitoring and eHealth solutions for assessing patients with chronic illnesses as diabetes, asthma and hypertension have previously shown great advantages in better disease control and improvement of symptoms. A similar eHealth solution for patients with RA is expected to be advantageous both for patients and the health care system.

The current trial is designed to assess if an eHealth solution for homebased disease activity monitoring is superior to the standard clinical disease monitoring strategy with respect to T2T goals. The main research question is whether the effectiveness of home-based disease activity monitoring via a home-based (eHealth) intervention is superior to standard clinical disease activity assessment in obtaining and maintaining a low(er) disease activity in patients with RA.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with rheumatoid arthritis
* Diagnosed with RA > 12 months
* Age between 18 and 85 years
* Computer and Internet connection at home and ability to employ these
* Hand function that allows self-testing of blood test at home.

Exclusion Criteria:

* Blood samples (creatinine, haemoglobin) outside lower normal limit - 5 % and upper normal limit + 5 % at screening.
* Blood samples (thrombocytes and leukocytes) outside lower normal limit - 15 % and upper normal limit + 15 % at screening
* Blood samples (ALT) outside lower normal limit - 100 % and upper normal limit + 100 % at screening
* Previously diagnosed with neutropenia and/or pancytopenia
* Dementia or other cognitive/physical deficiency that prevents participation
* Vision impairment that prevents the use of the devices and computer.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-08-18 (Actual); Primary Completion 2020-08-18 (Actual); Study Completion 2020-08-18 (Actual)

PRIMARY OUTCOMES:
Average DAS28-CRP over time | 6 months from baseline
  The Disease Activity Score (DAS) is a combined index that has been developed to measure the disease activity in patients with RA. It is a composite of standard clinical, laboratory data, and patient-reported data. The DAS28-CRP requires a standard blood sample (20 ml) to be drawn and analysed.

SECONDARY OUTCOMES:
DAS28-CRP<3.2 | 6 months from baseline
  Proportion of patients with low disease activity (LDA) defined as DAS28-CRP<3.2
DAS28-CRP<2.6 | 6 months from baseline
  Proportion of patients in remission defined as DAS28-CRP<2.6
Remission | 6 months from baseline
  Proportion of patients fulfilling the provisional and adapted ACR/EULAR remission criteria
The Short Form (36) Health Survey(The SF-36) | Change in the overall scores of the short form 36 questionnaire
  Change in the overall scores of the short form 36 questionnaire.
  The SF-36 is a patient-reported survey of patient health. It consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability.
Swollen-joint count, | 6 months from baseline
  Swollen-joint count, of 28 joints examined
Tender-joint count | 6 months from baseline
  Tender-joint count, of 28 joints examined
Physician's Global Assessment | 6 months from baseline
  Physician's Global Assessment - 0-100 mm VAS
Patient's Global Assessment | 6 months from baseline
  Patient's Global Assessment - 0-100 mm VAS
Patient's assessment of pain | 6 months from baseline
  Patient's assessment of pain - 0-100 mm VAS
HAQ-DI | 6 months from baseline
  HAQ-DI - score: 0-3
High-sensitivity C-reactive protein | 6 months from baseline
  High-sensitivity C-reactive protein - mg/L
Erythrocyte sedimentation | 6 months from baseline
  Erythrocyte sedimentation - mm/hr
Simplified Disease Activity Index | 6 months from baseline
  Simplified Disease Activity Index - score 0.1 to 86.0
Clinical Disease Activity Index | 6 months from baseline
  Clinical Disease Activity Index - score 0 to 76
Rheumatoid Arthritis Impact of Disease (RAID) | 6 months from baseline
  7 (NRS) questions assessed as a number between 0 and 10.
Brief illness perception questionnaire (IPQ-B) | 6 months from baseline
  Generic questionnaire developed to measure illness perception. The IPQ-B contains eight items and one causal scale. Items 1-8 are rated using a 0-to-10 response scale, item 9 is a memo field. Five of the items assess cognitive illness representations: consequences (Item 1), timeline (Item 2), personal control (Item 3), treatment control (Item 4), and identity (Item 5). Two of the items assess emotional representations: concern (Item 6) and emotions (Item 8). One item assesses illness comprehensibility (Item 7).
  A low score on items number 1,2,5,6 and 8 indicates that the illness is perceived as benign while a low score on the items 3, 4 and 7 indicates that the illness is perceived as threatening. By reversing these three items it is possible to compute an overall score. A higher score reflects a more threatening view of the illness.

CONTACTS AND LOCATIONS:
Overall Officials: Henning Bliddal, DMSc, Principal Investigator — The Parker Institute
Locations (2):
- Institute of Rheumatology, Charles University, Prague, Prague, Czechia
- The Parker Institute, Frederiksberg Hospital, Copenhagen, Denmark